CLINICAL TRIAL: NCT02890225
Title: Effect Of Renal Residual Stones c Treated By External Physical Vibration Lithecbole(EPVL) In m Different Time n After Retrograde Intrarenal w Surgery(RIRS):At y Multi-center z Prospective Randomized Controlled Trial
Brief Title: Comparison Of External Physical Vibration Lithecbole(EPVL) In Different Time After Retrograde Intrarenal Surgery(RIRS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Zhengzhou
Record Dates: First submitted 2016-08-25; First posted 2016-09-07 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Calculi
Keywords: stones; external physical vibration lithecbole
MeSH Terms: conditions — Calculi

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3 (Other): Patients in 3 days
  Interventions: Procedure: 3 days after
- 10 (Other): Patients in10ys
  Interventions: Procedure: 10days after
- 30 (Experimental): Patients in10ys
  Interventions: Procedure: EPVL performed in30days after RIRS

INTERVENTIONS:
Procedure: 3 days after — in 3 days after RIRS.
  Arms: 3
Procedure: 10days after — in10 days after RIRS.
  Arms: 10
Procedure: EPVL performed in30days after RIRS — Patients in Group C undergo EPVL in630days after RIRS.
  Arms: 30

SUMMARY:
The treatment of renal calculus by retrograde intrarenal surgery(RIRS) isn't able to eliminate stone completely

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of external physical vibration lithecbole for the treatment of residual stone in different time (3 days ,7 days and 14 days) after the operation of RIRS

ELIGIBILITY:
Inclusion Criteria:

1.Age of 18-75 years;

Exclusion Criteria:

1.Urinary tract anomalies, stricture or obstruction;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from stone free rate(SFR) with different follow-up periods | Patients in group A and group B return hospital respectively in 1,2 and 4 weeks after RIRS,patients in group C return hospital respectively in 2 and 4 weeks after RIRS.
  Primary SFR is assessed by abdominal plain film （KUB）in different follow-up periods after operation. Stone-free status are defined as either the absence of any residual stone fragments.

SECONDARY OUTCOMES:
Extracorporeal physical vibration complications | Patients in group A and group B return hospital respectively in 1,2 and 4 weeks after RIRS,patients in group C return hospital respectively in 2 and 4 weeks after RIRS.
  Complication is defined as any adverse event occurred

CONTACTS AND LOCATIONS:
Overall Officials: EB Wang, PH.D, Study Chair — Second Affiliated Hospital of Zhengzhou University
Locations (1):
- The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No